CLINICAL TRIAL: NCT03080428
Title: Prospective Multicenter Randomized Study Assessing Genomic Test Impact on Shared Decision of Adjuvant Chemotherapy in Patients With ER-positive, Her2-negative Early Breast Cancer With Uncertainty on the Indication of Chemotherapy Using Standard Assessments.
Brief Title: Assessment of Genomic Test Impact on Shared Decision of Adjuvant Chemotherapy in ER-positive, Her2-negative Early Breast Cancer
Acronym: OPTIGEN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study has been withdrawn because of lack of funding
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: UC-0140/1620; 2016-A01731-50 (Other: Id-RCB); UCBG 2-15 (Other: UNICANCER)
Record Dates: First submitted 2017-03-09; First posted 2017-03-15 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: ER-positive Her2-negative Early Breast Cancer
Keywords: Breast cancer; ER-positive; Her-2 negative; genomic test
MeSH Terms: conditions — Breast Neoplasms | interventions — Genetic Profile

STUDY DESIGN:
Intervention Model Description: Patients will be identified prior to surgery based on biopsy results. During the post-operative multidisciplinary decision-making meeting, a first therapeutic decision to prescribe or not an adjuvant chemotherapy will be taken according to usual clinical and histopathological markers and official guidelines in use in the center. After the patient has signed the inform consent form, the surgical sample will be sent by the investigator site to a selected genomic platform according to the randomization result.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Endopredict® (Active Comparator): genomic test Endopredict® realized on surgery tumour samples
  Interventions: Diagnostic Test: Genomic test
- Prosigna® (Active Comparator): genomic test Prosigna® realized on surgery tumour samples
  Interventions: Diagnostic Test: Genomic test
- OncotypeDX® (Active Comparator): genomic test OncotypeDX® realized on surgery tumour samples
  Interventions: Diagnostic Test: Genomic test
- Mammaprint® assay (Active Comparator): genomic test Mammaprint® assay realized on surgery tumour samples
  Interventions: Diagnostic Test: Genomic test

INTERVENTIONS:
Diagnostic Test: Genomic test — genomic test realized on surgery block or formalin-fixed paraffin-embedded slides

SUMMARY:
The need/benefit of adjuvant chemotherapy could be negligible for a certain category of patient with newly diagnosed unilateral non metastatic breast cancer. Physicians are sometimes divided between the administration of adjuvant treatment and no administration when the risk of distant relapse at 10 years is around 10% with uncertainty and a theoretical benefit of chemotherapy is less than 5% at 10 years according to guidelines in use in the center.

Several genomic tests have been developed this last decade. These tests use a sample of breast cancer tissue to analyze the activity of a group of genes. Knowing whether certain genes are present or absent, overly active or not active enough, can help physicians predict the risk of recurrence.

In addition to standard pathological characteristics, a genomic test could be helpful in making treatment decisions, such as whether or not chemotherapy should be part of the treatment plan. First generation prognostic tests are currently widely used worldwide to guide decision making regarding adjuvant chemotherapy (OncotypeDX™ Mammaprint®). Prognostic tests have reached a level of evidence 1A, with the results of the prospective randomized trial "Mindact". In the "Mindact" trial, among women with early-stage breast cancer who were at high clinical risk and low genomic risk for recurrence, the receipt of no chemotherapy on the basis of the 70-gene signature led to a 5-year rate of survival without distant metastasis that was 1.5 percentage points lower than the rate with chemotherapy. Given these findings, approximately 46% of women with breast cancer who are at high clinical risk might not require chemotherapy. The health-economic value of such signatures in the general population of patients with localized breast cancer appears very low at current costs.

Meanwhile, next generation prognostic signatures have been developed that have integrated clinical parameters and suggest high added value beyond all standard and traditional characteristics including tumor burden, grade, Estrogen Receptor (ER) and Progesterone Receptor (PR), Her2, age and also standard assessment of proliferation.

In this study, the clinical utility of genomic tests (Endopredict®, Prosigna®, OncotypeDX®, Mammaprint® assay) defined as impact on chemotherapy decision in the adjuvant setting in patients with ER-positive, Her2-negative early breast cancer with uncertainty on the indication of chemotherapy using standard assessments will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Woman, Age ≥ 18 years;
2. Performance status 0 or 1 (according to World Health Organization criteria);
3. Patient with newly diagnosed, unilateral, localized, histologically confirmed, invasive breast cancer; Note: Multicentric/multifocal tumors are allowed provided a maximum of 3 lesions are present, and all are ER > 10% or Allred ≥ 4, Her2-negative (genomic test will be performed on the lesion considered the most pertinent by the multidisciplinary team)
4. Fully operated breast cancer including complete resection of breast tumor and adequate axillary surgery;
5. Available surgical material (formalin-fixed, paraffin-embedded) for genomic test evaluation;
6. ER-positive by immuno-histochemical (>10% cells stained or Allred Score≥4);
7. HER2-negative by IHC (score 0 or 1+) and/or fluorescence in situ hybridization/silver in situ hybridization/chemiluminescent in situ hybridization ;
8. Uncertainty regarding the toxicity/benefit of adjuvant chemotherapy, outlined in the following situations:

   * Grade 1: pT3 or 1-3 node positive
   * Grade 2: pT1 pN0 but high proliferation (Ki67 >20%) or lympho-vascular emboli, or 1-3 node positive
   * Grade 2 : pT2 pN0
   * Grade 3: pT1 pN0
9. Adequate renal, hepatic, cardiac and hematopoietic functions for a chemotherapy administration;
10. Willingness and ability to comply with scheduled visits as well as with test results and chemotherapy decision according to the latest;
11. Signed informed consent and Health insurance coverage.

Exclusion Criteria:

1. Non operable, bilateral, locally advanced, T4 or metastatic breast cancer;
2. HER2 Overexpression, as assessed by 3+ IHC or FISH/SISH/CISH amplification;
3. Diagnosis of any previous malignancy within the last 5 years, except for adequately treated basal cell carcinoma, or squamous cell skin carcinoma, or in situ cervical carcinoma;
4. Any previous systemic or locoregional treatment for the present breast cancer;
5. Documented inherited predisposition with BRCA1/2 or TP53 mutation;
6. Previous hormone replacement therapy (HRT) stopped less than 2 weeks before surgery;
7. Previous treatment for the present breast cancer;
8. Person unable to give informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of genomic tests clinical utility | At the end of the inclusion period: 12 months
  Pairwise comparisons between genomic tests in terms of percentage of changes between initial adjuvant chemotherapy decision and final receipt of chemotherapy (yes/no)

SECONDARY OUTCOMES:
Distant disease-free survival in patients who do not receive chemotherapy | 5 years
  5-year distant disease-free survival among the pooled cohort of patients who did not receive chemotherapy
Distant disease-free survival in patients who do not receive chemotherapy based on genomic test result. | 5 years
  5-year distant disease-free survival in patients who did not receive chemotherapy based on genomic test result
Reason for discordant final decision when they occur | 12 months
  Number of decision changes according to the test results. Physicians' and patients' reasons for "non-compliance" with the test's results will be recorded (a threshold at 10% 10 year distant recurrence risk will be chosen)
Feasibility of test in terms of time interval. | 12 months
  Time interval between prescription and result of the test (% < 10 days)
differences in results between local and central reading of ER, PR, Her2 and Ki67 | 12 months
  A comparison with local evaluation of HR, Her2, and ki-67 will be made
Change of therapy based on the genomic test findings in a virtual tumour board | 12 months
  Choice of therapy in a virtual tumour board based on the genomic test findings
Evaluation of the cost effectiveness of genomic tests | 5 years
  Medico-economic impact based on results of the "Optisoin 01" study

CONTACTS AND LOCATIONS:
Overall Officials: Roman Rouzier, MD, Principal Investigator — Institut Curie

IPD SHARING:
Plan to Share IPD: Undecided